CLINICAL TRIAL: NCT05574153
Title: Metabolic Risk Factors and Myocardial Oxygenation Reserve (META-MORE)
Brief Title: Metabolic Risk Factors and Myocardial Oxygenation Reserve
Acronym: (META-MORE)
Status: Recruiting | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Matthias Friedrich, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2021-7267
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Metabolic Syndrome
Keywords: Myocardial oxygenation
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patient Participant: Participants with known Metabolic Syndrome (MetS)
  Interventions: Diagnostic Test: Cardiac MRI
- Healthy Volunteers: NonS-moking participants with no known pre-existing conditions and who do not take any medications
  Interventions: Diagnostic Test: Cardiac MRI

INTERVENTIONS:
Diagnostic Test: Cardiac MRI — Participants will undergo an oxygenation-sensitive cardiac MRI and, during the scan, perform a vasoactive breathing maneuver composed of a period of paced hyperventilation followed by a voluntary maximal breath hold.
  Other Names: Breathing Maneuvers

SUMMARY:
The purpose of this study is to use MRI images using the OS-CMR technique to view the differences in the hearts of healthy volunteers and participants with a condition called Metabolic Syndrome. The objectives of this project are to compare these two groups and to view how health risks, blood test results, and the time since a Metabolic diagnosis can affect heart health.

DETAILED DESCRIPTION:
Myocardial oxygenation changes during vasoactive breathing maneuvers, observed with oxygenation-sensitive cardiac MRI, will be identified and compared between individuals considered healthy and those fitting the criteria of the Metabolic Syndrome.

ELIGIBILITY:
Inclusion Criteria:

Patient Participants:

* Age 18-80
* Informed Consent
* Diagnosis of MetS (through at least 3 MetS characteristics (abdominal obesity, high triglyceride level, low HDL cholesterol, high systolic blood pressure, and high fasting glucose levels)

Healthy Volunteers:

* Age 18-80
* No known current or pre-existing significant medical problems that would affect the cardiovascular or respiratory system
* No Smoking

Exclusion Criteria:

* General MRI contraindications*
* Pacemakers, defibrillating wires, implanted defibrillators, intracranial aneurysm clips, metallic foreign bodies in the eyes, knowledge or suspicion of pregnancy.
* Consumption of caffeine (coffee, tea, cocoa, chocolate, "energy drink") during the 12 hours prior to the exam

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be composed of participants with known MetS, based on the identified risk factors, and healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Global and segmental Myocardial oxygenation reserve (MORE) | Baseline
  A t-test will be used to assess the difference in global and segmental MORE, at rest, during hyperventilation, and throughout breath hold, between healthy and volunteers and MetS patients.
Relation between Breathing maneuver induced MORE and known MetS risk factors. | Baseline
  A linear regression will assess the relation between Breathing maneuver induced MORE and known MetS risk factors, biomarkers, and time since diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- The Reseach Institute of the McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No